CLINICAL TRIAL: NCT05072665
Title: EFFECT OF FOOD ALLERGENS ON DUODENAL MUCOSAUS BY CONFOCAL ENDOSCOPIC IMAGING Cellvizio
Brief Title: Fast Allergy Sensitivity Test
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Trocadéro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01267-34
Record Dates: First submitted 2021-09-01; First posted 2021-10-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATIENT WITH Irritable Bowel Syndrome (Experimental): 2.5 ml of 10% fluorescein (SERB) will be administered to the patient intravenously. after the fluorescein injection.
  A first food allergen will be applied to the duodenal mucosa starting with the most distal part of the duodenum. After 2 minutes following the application of the allergen, observation using the endomicroscopy system can begin by applying the GastroFlex ™ UHD probe to the duodenal mucosa where the allergen has been projected. . Observation will last up to 3 minutes per site observed. If no reaction is observed, the same manipulation will be carried out using a new allergen. If the observed reaction is positive, the test will be stopped
  Interventions: Device: HIGH ECHOENDOSCOPY WITH THE FAST PROCEDURE

INTERVENTIONS:
Device: HIGH ECHOENDOSCOPY WITH THE FAST PROCEDURE — HIGH ECHOENDOSCOPY WITH THE FAST PROCEDURE

SUMMARY:
Irritable Bowel Syndrome (IBS), or functional colopathy, is a chronic disease that affects 10% to 20% of the world's population.This syndrome is characterized by chronic abdominal pain or discomfort as well as a change in bowel habits (constipation or diarrhea) in the absence of structural or metabolic abnormalities (e.g. celiac disease, Crohn's disease). These symptoms have an impact on the quality of life of these patients who must therefore integrate the management of their disease into their daily life.IBS is subdivided into 3 subtypes according to the predominant symptom: the IBS-D subtype which groups together patients who have a predominance of diarrheal episodes, the IBS-C subtype which groups together patients who have a predominance of '' episodes of constipation and finally the IBS-M subtype which includes patients whose two symptoms mentioned above are observed without predominance

DETAILED DESCRIPTION:
In 2014, Fritscher-Ravens et al., Described for the first time the value of endomicroscopy in the diagnosis of food allergies by observing the reaction of the duodenal mucosa to food allergens in patients with IBS. They assessed the structural and functional changes that were occurring in the intestinal lining in vivo and noted the following changes at the cellular level:

* The layers of epithelial cells break down and are removed forming voids and inducing an immediate increase in the fluid permeability of the duodenal mucosa. As a result, the contrast agent penetrates the lumen, widening the space between the villi and changing the appearance from black to white.
* These changes were usually seen between 2 min and 4 min after exposure to the allergen.

This procedure, called FAST (Food Allergy Sensitivity Test), has since been used routinely in certain centers in Germany. However, few studies have been published that have shown the reproducibility of these results as well as the performance of this new test. The study that the investigators propose to conduct is a prospective multicenter pilot study conducted in the Trocadero Clinic

1. Pre-test consultation The patients will first be seen by a nutritionist. During this consultation, eligible patients will be offered, in addition to endoscopy performed in current practice, the possibility of performing the FAST test during endoscopy. Up to 7 days before the operation, a questionnaire allowing the assessment of the severity of symptoms (IBS-SSS) will be provided to the patient who has agreed to participate in the study. The answers to the questionnaire will be used as a reference to assess the evolution of symptoms if a food exclusion diet were to be put in place following the procedure. Finally, two to three days before the FAST test, the patient will be asked to follow an exclusion diet and consume only hypoallergenic nutritional foods: rice, potatoes, olive oil, salt.

2 Carrying out the test Before the start of the test, a standard high-end endoscopy will be performed to look for any signs of structural mucosal abnormalities that suggest gastrointestinal disease. In the event of a mucosal abnormality observed on endoscopy, the CLE FAST procedure will be canceled. In the case of mild reflux disease, the test may be done.

Prior to the first challenge, 2.5 ml of 10% fluorescein (SERB) will be administered to the patient intravenously.

Before any challenge and after the fluorescein injection, to establish a comparison image, a first acquisition with the endomicroscopy system of the duodenal mucosa will be carried out on a minimum of 4 sites (approximately 20 seconds each) to verify the integrity of the mucosa.

During the acquisition of the reference sequences and during all subsequent acquisitions, areas of the mucosa that show bleeding and other visible signs of inflammation will not be imaged in order to avoid false positives.

Once the reference images have been acquired, a first food allergen will be applied to the duodenal mucosa starting with the most distal part of the duodenum. After 2 minutes following the application of the allergen, observation using the endomicroscopy system can begin by applying the GastroFlex ™ UHD probe to the duodenal mucosa where the allergen has been projected. . Observation will last up to 3 minutes per site observed. If no reaction is observed, the same manipulation will be carried out using a new allergen. If the observed reaction is positive, the test will be stopped.

The test can be performed using up to 5 different allergens as long as the total time after fluorescein injection does not exceed 30min.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosis of irritable bowel syndrome according to the ROME IV classification
* Negative blood test: determination of IgE; anti-transglutaminase IgA assay (celiac disease)
* Symptoms potentially related to a food allergy
* Sufficient cooperation and understanding to comply with the requirements of the study with a post-Cellvizio medical examination at 2 weeks, 2 months and 6 months

Exclusion Criteria:

* Patients under 18
* Patient benefiting from a legal protection measure (curatorship, guardianship, etc.)
* Pregnant or breastfeeding woman
* Known allergy to fluorescein
* Digestive cancer (stomach cancer colon rectal cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Observation, at the time of the endomicroscopy procedure, of ruptures / leaks in the mucous membranes and intercellular extravasation of plasma fluid labeled with fluorescein in the intercellular space | day 1
SCORE ROME IV | DAYS 28
  QUESTIONNARY
SCORE ROME IV | 2 months
  QUESTIONNARY
SCORE ROME IV | 6 months
  QUESTIONNARY

SECONDARY OUTCOMES:
SCORE OBS-SSS | days 28
  QUESTIONNARY
SCORE OBS-SSS | 2months
  QUESTIONNARY
SCORE OBS-SSS | 6 months
  QUESTIONNARY
RESULT OH THE DIET | 6 MONTHS
  consultation

CONTACTS AND LOCATIONS:
Locations (1):
- clinique du Trocadero, Paris, France

IPD SHARING:
Plan to Share IPD: No